CLINICAL TRIAL: NCT01770340
Title: Nerve Grafting With an Allograft During Radical Prostatectomy - Extended Follow-up in a Prospective Randomized Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment, Interim analysis: The rates of pts who reached primary and secondary endpoints were lower than expected.
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-ZH-NR:2010-0004/0
Record Dates: First submitted 2012-12-13; First posted 2013-01-17 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
Keywords: radical prostatectomy; erectile function; nerve grafting; allogenic; prostate cancer; Allogenic nerve graft; Time required for nerve grafting
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Sham Comparator): Radical prostatectomy without implantation of allograft
  Interventions: Procedure: Radical prostatectomy without implantation of allograft
- Treatment group (Experimental): Radical prostatectomy with implantation of allograft
  Interventions: Biological: Radical prostatectomy with implantation of allograft

INTERVENTIONS:
Biological: Radical prostatectomy with implantation of allograft — Interposition of resected neurovascular bundles with allograft Avance®
  Arms: Treatment group
Procedure: Radical prostatectomy without implantation of allograft — No interposition of resected neurvascular bundles
  Arms: Control group

SUMMARY:
Earlier studies were able to show that an improvement of the erectile function following a non-nerve sparing radical prostatectomy could be achieved using an autologous nerve graft.

The investigators evaluate the use of the implantation of the allogenic nerve graft Avance® in patients undergoing non nerve-sparing radical prostatectomy.

DETAILED DESCRIPTION:
In this prospective randomised and single-blind, clinical phase-IV study, 60 patients are randomized into the treatment group and the control group. The follow-up is at least 24 months.

The inclusion criteria were localized prostate cancers cT3 and/or Gleason score ≥ 7 (a or b) and/or prostate-specific antigen (PSA) ≥ 20 ng/ml and furthermore an erectile function with an IIEF ≥ 21 (IIEF-6).

The operation carried out is a standardised, robot assisted laparoscopic radical prostatectomy with total excision of both neurovascular bundles.

The Outcome measurement is done with the "quality of life questionnaire before and after prostate surgery" that includes the "International Index of Erectile Function" (IIEF) questionnaire.

The limitations are a small cohort, a short observation period and the lack of statistical analysis due to a still low number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Localized intermediate-risk or high-risk prostate cancer cT3
* Gleason score ≥ 7 (3+4 and/or 4+3) and/or
* PSA ≥ 20 ng/ml
* intact preoperative erectile function with an IIEF ≥ 21 (IIEF-6).

Exclusion Criteria:

* IIEF < 21
* Operations in the past 6 months which could limit the erectile function
* Erectile dysfunction in the history or current medication for erectile dysfunction
* Current involvement in another comparable study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2017-04 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Erectile function score (IIEF: international index of erectile function) after non nerve sparing radical prostatectomy | 24 months
  Erectile function score (IIEF: international index of erectile function) after non nerve sparing radical prostatectomy. To show a complete impotence in the control group and an enhancement of the initial postoperative impotence in the treatment group

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 months
  Monitoring of side effects and complications in connection with the nerve-implantation.

OTHER OUTCOMES:
Documented will be the extra time required for the nerve implantation | at the time of operation
  How much operation-time takes the nerve implantation? The time is stopped which is required for the implantation of the nerve. Start is when the prostate was removed and was deposited in the extraction bag. Stop when the anastomosis of the nerves is stitched and the anastomosis of the urethra begins.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert John, Chefarzt, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland